CLINICAL TRIAL: NCT01877187
Title: Lipiodol as an Imaging Biomarker of Tumor Necrosis After Transcatheter Chemoembolization Therapy in Patients With Primary and Metastatic Liver Cancer
Brief Title: Lipiodol as an Imaging Biomarker in Patients With Primary and Metastatic Liver Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: J12115; NA_00074005 (Other: Johns Hopkins Institutional Review Board); HIC1601017054 (Other: Yale University)
Record Dates: First submitted 2013-03-27; First posted 2013-06-13 (Estimated); Results first posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Liver Cancer
Keywords: Primary liver cancer; Metastatic liver cancer
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Ethiodized Oil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lipiodol (Other): Lipiodol, 10cc per TACE.
  Interventions: Drug: Lipiodol

INTERVENTIONS:
Drug: Lipiodol — Lipiodol is used as a carrier for chemotherapy agents and also as an occlusion agent. In TACE procedures, Lipiodol is mixed with the chemotherapy agent(s) and delivered to the tumor via the hepatic artery, causing necrosis of the targeted tumor(s).
  Other Names: Ethiodol

SUMMARY:
The purpose of this study is to determine the whether Lipiodol can be used as an imaging biomarker, predicting tumor response to therapy in patients with primary and metastatic liver cancer. Lipiodol-based transarterial chemoembolization (TACE) has been an accepted standard of care procedure for unresectable liver lesions for several decades. Lipiodol is used as a carrier for chemotherapy agents and also as an occlusion agent. In TACE procedures, Lipiodol is mixed with the chemotherapy agent(s) and delivered to the tumor via the hepatic artery, causing necrosis of the targeted tumor(s). Response to therapy will be evaluated every 1, 3 and 6 months by clinic visits, MRI/CT/PET scans and blood tests (to include assessment of liver function and tumor markers).

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older.
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2.
3. Childs class of A or B (up to 9).
4. Hepatocellular carcinoma (HCC) is unresectable with liver-predominant disease or subject has HCC and refused surgery or subject is diagnosed hepatic metastases from any solid tumor. (Multifocal HCC is acceptable, no diffuse HCC).
5. Subject is voluntarily participating in the study and has signed the informed consent.

Exclusion Criteria:

1. Contraindications to doxorubicin, cisplatin, or mytomycin-c administration (or specific mixture of chemotherapy drugs to be used).
2. Evidence of severe or uncontrolled systemic diseases.
3. Congestive cardiac failure >NYHA class 2 MI within 6 months, active coronary artery disease, cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers or digoxin, unstable angina, or laboratory finding that in the view of the investigator makes it undesirable for the patient to participate in the trial.
4. Known allergy to Lipiodol (Ethiodol), poppy seed oil, or iodinated contrast agents (that cannot be adequately mitigated with pre-procedure medication).
5. Main portal vein thrombosis is excluded; segmental or branch portal vein thrombosis is acceptable.
6. Subject is breastfeeding.
7. Subject is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Todd Schlachter, MD, Principal Investigator — Yale University
Locations (2):
- United States (2):
  - Smilow Cancer Center, New Haven, Connecticut
  - The Johns Hopkins Hospital, Baltimore, Maryland

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lipiodol
Started | 39 (21 HCC, 18 non-HCC)
Completed 30 Day f/u | 35 (18 HCC, 17 non-HCC)
Completed 90 Day f/u | 20 (11 HCC, 9 non-HCC)
Completed (Completed 180 day f/u) | 17 (10 HCC, 7 non-HCC)
Not Completed | 22
Not completed — Death | 2
Not completed — Withdrawal by Subject | 4
Not completed — Lost to Follow-up | 3
Not completed — Declining clinical status | 11
Not completed — Liver transplant | 2

BASELINE CHARACTERISTICS:
Arm/Group | Lipiodol
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.28 (10.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 23
  African American | 10
  Hispanic | 1
  Other | 5
Region of Enrollment [Number; unit: participants]
  United States | 39
Tumor Type [Count of Participants; unit: Participants]
  Hepatocellular carcinoma | 22
  Neuroendocrine: GI | 4
  Neuroendocrine: pancreatic | 2
  Neuroendocrine: bronchial | 1
  Cholangiocarcinoma | 8
  Cutaneous melanoma | 1
  Uveal melanoma | 1

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response by Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Lipiodol deposition in the tumor will be measured using non contrast CT. The images from the non contrast CT will also be correlated with RECIST response separately using contrast CT, MRI and PET imaging. Response rates taken at 30 days, 90 days, 180 days. Per Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI:
  Complete Response (CR): Disappearance of all target lesions Partial Response (PR): >= 30% decrease in the sum of the longest diameter of target lesions
  Overall Response (OR) = CR + PR
Time Frame: 30 days, 90 days, and 180 days
Population: 18 HCC and 16 non-HCC subjects had complete data for analysis at 30day f/u, 11 HCC and 7 non-HCC at 90 day f/u, and 11 HCC and 5 non-HCC at 180 day f/u.
Measure: Count of Participants; unit: Participants
Groups:
- Lipiodol (HCC); Lipiodol (Non-HCC): Lipiodol, 10cc per TACE.
  Lipiodol: Lipiodol is used as a carrier for chemotherapy agents and also as an occlusion agent. In TACE procedures, Lipiodol is mixed with the chemotherapy agent(s) and delivered to the tumor via the hepatic artery, causing necrosis of the targeted tumor(s).
Arm/Group | Lipiodol (HCC) | Lipiodol (Non-HCC)
Number analyzed (Participants) | 18 | 16
Participants
  30 day f/u: Responders | 1 | 1
  30 day f/u: Non-responders | 17 | 15
  90 day f/u: number analyzed (Participants) | 11 | 7
  90 day f/u: Responders | 5 | 3
  90 day f/u: Non-responders | 6 | 4
  180 day f/u: number analyzed (Participants) | 11 | 5
  180 day f/u: Responders | 4 | 2
  180 day f/u: Non-responders | 7 | 3

2. Primary Outcome: Baseline Enhancing Tumor and Response by RECIST Criteria
Description: Analysis of enhancing tumor (% of tumor that arterially enhances on MRI imaging) to correlate with responders/nonresponders by RECIST criteria. Responders are subjects that demonstrated Complete Response or Partial Response by RECIST criteria. Nonresponders are all other subjects.
Time Frame: 30 days, 90 days, 180 days
Population: 16 HCC and 14 non-HCC subjects had applicable data for analysis at 30day f/u, 9 HCC and 6 non-HCC at 90 day f/u, and 9 HCC and 4 non-HCC at 180 day f/u.
Measure: Median (Full Range); unit: % tumor enhancement
Groups:
- Overall: Combined Lipiodol (HCC) and Lipiodol (Non-HCC)
Arm/Group | Lipiodol (HCC) | Lipiodol (Non-HCC) | Overall
Number analyzed (Participants) | 16 | 14 | 30
% tumor enhancement
  (30 day) Responders: number analyzed (Participants) | 1 | 1 | 2
  (30 day) Responders | 95.1 [95.1 to 95.1] | 97.30 [97.3 to 97.3] | 96.2 [95.1 to 97.3]
  (30 day) Nonresponders: number analyzed (Participants) | 15 | 13 | 28
  (30 day) Nonresponders | 53.4 [6.1 to 99.8] | 50.7 [6.0 to 81.9] | 52.1 [6.0 to 99.8]
  (90 day) Responders: number analyzed (Participants) | 4 | 2 | 6
  (90 day) Responders | 65.2 [29.6 to 99.8] | 89.6 [81.9 to 97.3] | 79.4 [29.6 to 99.8]
  (90 day) Nonresponders: number analyzed (Participants) | 5 | 4 | 9
  (90 day) Nonresponders | 50.6 [36.3 to 93.4] | 30.4 [6.0 to 67.8] | 42.4 [6.0 to 93.4]
  (180 day) Responders: number analyzed (Participants) | 3 | 2 | 5
  (180 day) Responders | 77.0 [53.4 to 99.8] | 89.6 [81.9 to 97.3] | 81.9 [53.4 to 99.8]
  (180 day) Nonresponders: number analyzed (Participants) | 6 | 2 | 8
  (180 day) Nonresponders | 46.2 [29.6 to 93.4] | 43.1 [18.4 to 67.8] | 46.2 [18.4 to 93.4]
Statistical Analysis 1: Comparison: Overall; Sample size of 60 achieves 80% power to detect a Pearson correlation coefficient of 0.35 with a two-sided significant level of 0.05. Sample size of 30 will allow for detecting a Pearson correlation coefficient of 0.49 in each subgroup; Test type: Other; p = .06, Wilcoxon (Mann-Whitney) — Statistical significance defined as p <= .05. Result is for Day 30 timepoint
Statistical Analysis 2: Comparison: Overall; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = .09, Wilcoxon (Mann-Whitney) — Statistical significance defined as p <= 0.05. Data for 90 day timepoint
Statistical Analysis 3: Comparison: Overall; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.034, Wilcoxon (Mann-Whitney) — Statistical significance defined as p <= 0.05. Data for 180 day timepoint

3. Secondary Outcome: Tumor Response by Modified Response Evaluation Criteria in Solid Tumors (mRECIST)
Description: Lipiodol deposition in the tumor will be measured using non contrast CT. The images from the non contrast CT will also be correlated with mRECIST response separately using contrast CT, MRI and PET imaging. Response rates taken at 30 days, 90 days, 180 days. Per modified Response Evaluation Criteria in Solid Tumors (mRECIST):
  Complete Response (CR): Disappearance of all intratumoral arterial enhancement in target lesions Partial Response (PR): At least 30% decrease in the sum of the diameters of viable (enhancement in the arterial phase) target lesions Overall Response (OR) = CR + PR
Time Frame: 30 days, 90 days, and 180 days
Population: 18 HCC and 14 non-HCC subjects had complete data for analysis at 30day f/u, 11 HCC and 7 non-HCC at 90 day f/u, and 11 HCC and 5 non-HCC at 180 day f/u.
Measure: Count of Participants; unit: Participants
Arm/Group | Lipiodol (HCC) | Lipiodol (Non-HCC)
Number analyzed (Participants) | 18 | 14
Participants
  30 day f/u: Responders | 9 | 2
  30 day f/u: Non-responders | 9 | 12
  90 day f/u: number analyzed (Participants) | 11 | 7
  90 day f/u: Responders | 6 | 3
  90 day f/u: Non-responders | 5 | 4
  180 day f/u: number analyzed (Participants) | 11 | 5
  180 day f/u: Responders | 6 | 2
  180 day f/u: Non-responders | 5 | 3

4. Secondary Outcome: Baseline Enhancing Tumor and Response by mRECIST Criteria
Description: Analysis of enhancing tumor (% of tumor that arterially enhances on MRI imaging) to correlate with responders/nonresponders by mRECIST criteria. Responders are subjects that demonstrated Complete Response or Partial Response by mRECIST criteria. Nonresponders are all other subjects.
Time Frame: 30 days, 90 days, 180 days
Population: as for outcome 2
Measure: Median (Full Range); unit: % tumor enhancement
Arm/Group | Lipiodol (HCC) | Lipiodol (Non-HCC) | Overall
Number analyzed (Participants) | 16 | 14 | 30
% tumor enhancement
  (30 day) Responders: number analyzed (Participants) | 7 | 2 | 9
  (30 day) Responders | 95.1 [6.1 to 99.8] | 53.7 [29.2 to 78.2] | 78.2 [6.1 to 99.8]
  (30 days) Nonresponders: number analyzed (Participants) | 9 | 12 | 21
  (30 days) Nonresponders | 50.6 [9.6 to 93.4] | 52.7 [6.0 to 97.3] | 50.7 [6.0 to 97.3]
  (90 days) Responders: number analyzed (Participants) | 4 | 2 | 6
  (90 days) Responders | 74.1 [53.4 to 99.8] | 89.6 [81.9 to 97.3] | 79.4 [53.4 to 99.8]
  (90 days) Nonresponders: number analyzed (Participants) | 5 | 4 | 9
  (90 days) Nonresponders | 41.8 [29.3 to 93.4] | 30.4 [6.0 to 67.8] | 41.8 [6.0 to 93.4]
  (180 days) Responders: number analyzed (Participants) | 4 | 2 | 6
  (180 days) Responders | 74.1 [29.6 to 99.8] | 50.1 [18.4 to 81.9] | 74.1 [18.4 to 99.8]
  (180 days) Nonresponders: number analyzed (Participants) | 5 | 2 | 7
  (180 days) Nonresponders | 50.6 [36.3 to 93.4] | 82.5 [67.8 to 97.3] | 53.4 [36.3 to 97.3]
Statistical Analysis 1: Comparison: Overall; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.19, Wilcoxon (Mann-Whitney) — Statistical significance defined as p <= 0.05. Data for 30 day timepoint
Statistical Analysis 2: Comparison: Overall; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.011, Wilcoxon (Mann-Whitney) — Statistical significance defined as p <= 0.05. Data for 90 day timepoint
Statistical Analysis 3: Comparison: Overall; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.94, Wilcoxon (Mann-Whitney) — Statistical significance defined as p <= 0.05. Data for 180 day timepoint

5. Secondary Outcome: Tumor Response by World Health Organization (WHO) Criteria
Description: Lipiodol deposition in the tumor will be measured using non contrast CT. The images from the non contrast CT will also be correlated with WHO response separately using contrast CT, MRI and PET imaging. Response rates taken at 30 days, 90 days, 180 days. Per WHO criteria:
  Complete Response (CR): disappearance of all lesions for >= 4 weeks. Partial Response (PR): At least 50% decrease in sum of the products of diameters of target lesions.
  Overall Response: CR + PR.
Time Frame: 6 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Lipiodol (HCC) | Lipiodol (Non-HCC)
Number analyzed (Participants) | 18 | 16
Participants
  30 day f/u: Responders | 2 | 1
  30 day f/u: Non-responders | 16 | 15
  90 day f/u: number analyzed (Participants) | 11 | 7
  90 day f/u: Responders | 4 | 3
  90 day f/u: Non-responders | 7 | 4
  180 day f/u: number analyzed (Participants) | 11 | 5
  180 day f/u: Responders | 4 | 2
  180 day f/u: Non-responders | 7 | 3

6. Secondary Outcome: Baseline Enhancing Tumor and Response by WHO Criteria
Description: Analysis of enhancing tumor (% of tumor that arterially enhances on MRI imaging) to correlate with responders/nonresponders by WHO criteria. Responders are subjects that demonstrated Complete Response or Partial Response by WHO criteria. Nonresponders are all other subjects.
Time Frame: 30 days, 90 days, 180 days
Population: as for outcome 2
Measure: Median (Full Range); unit: % tumor enhancement
Arm/Group | Lipiodol (HCC) | Lipiodol (Non-HCC) | Overall
Number analyzed (Participants) | 16 | 14 | 30
% tumor enhancement
  (30 day) Responders: number analyzed (Participants) | 1 | 1 | 2
  (30 day) Responders | 95.1 [95.1 to 9.51] | 97.3 [97.3 to 97.3] | 96.2 [95.1 to 97.3]
  (30 days) Nonresponders: number analyzed (Participants) | 15 | 13 | 28
  (30 days) Nonresponders | 53.4 [6.1 to 99.8] | 50.7 [6.0 to 81.9] | 52.1 [6.0 to 99.8]
  (90 days) Responders: number analyzed (Participants) | 3 | 2 | 5
  (90 days) Responders | 77.0 [53.4 to 99.8] | 89.6 [81.9 to 97.3] | 81.9 [53.4 to 99.8]
  (90 days) Nonresponders: number analyzed (Participants) | 6 | 4 | 10
  (90 days) Nonresponders | 46.2 [29.6 to 93.4] | 30.4 [6.0 to 67.8] | 42.1 [6.0 to 93.4]
  (180 days) Responders: number analyzed (Participants) | 3 | 1 | 4
  (180 days) Responders | 77.0 [53.4 to 99.8] | 97.3 [97.3 to 97.3] | 87.5 [53.4 to 99.8]
  (180 days) Nonresponders: number analyzed (Participants) | 6 | 3 | 9
  (180 days) Nonresponders | 46.2 [29.6 to 93.4] | 67.8 [18.4 to 81.9] | 50.6 [18.4 to 93.4]
Statistical Analysis 1: Comparison: Overall; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.06, Wilcoxon (Mann-Whitney) — Statistical significance defined as p <= 0.05. Data for 30 day timepoint
Statistical Analysis 2: Comparison: Overall; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.017, Wilcoxon (Mann-Whitney) — Statistical significance defined as p <= 0.05. Data for 90 day timepoint
Statistical Analysis 3: Comparison: Overall; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.08, Wilcoxon (Mann-Whitney) — Statistical significance defined as p <= 0.05. Data for 90 day timepoint

7. Secondary Outcome: Tumor Response by European Association for the Study of the Liver (EASL) Criteria
Description: Lipiodol deposition in the tumor will be measured using non contrast CT. The images from the non contrast CT will also be correlated with EASL response separately using contrast CT, MRI and PET imaging. Response rates taken at 30 days, 90 days, 180 days. Per EASL response:
  Complete Response (CR): complete disappearance of enhancing tissue in target lesions Partial Response (PR): At least 50% decrease in area of enhancing tissue in target lesions.
  Overall Response: CR+PR
Time Frame: 6 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Lipiodol (HCC) | Lipiodol (Non-HCC)
Number analyzed (Participants) | 18 | 14
Participants
  30 day f/u: Responders | 11 | 2
  30 day f/u: Non-responders | 7 | 12
  90 day f/u: number analyzed (Participants) | 11 | 7
  90 day f/u: Responders | 7 | 5
  90 day f/u: Non-responders | 4 | 2
  180 day f/u: number analyzed (Participants) | 11 | 5
  180 day f/u: Responders | 7 | 4
  180 day f/u: Non-responders | 4 | 1

8. Secondary Outcome: Baseline Enhancing Tumor and Response by EASL Criteria
Description: Analysis of enhancing tumor (% of tumor that arterially enhances on MRI imaging) to correlate with responders/nonresponders by EASL criteria. Responders are subjects that demonstrated Complete Response or Partial Response by EASL criteria. Nonresponders are all other subjects.
Time Frame: 30 days, 90 days, 180 days
Population: as for outcome 2
Measure: Median (Full Range); unit: % tumor enhancement
Arm/Group | Lipiodol (HCC) | Lipiodol (Non-HCC) | Overall
Number analyzed (Participants) | 16 | 14 | 30
% tumor enhancement
  (30 day) Responders: number analyzed (Participants) | 9 | 2 | 11
  (30 day) Responders | 77.0 [6.1 to 99.8] | 87.8 [78.2 to 97.3] | 78.2 [6.1 to 99.8]
  (30 days) Nonresponders: number analyzed (Participants) | 7 | 12 | 19
  (30 days) Nonresponders | 50.1 [9.6 to 93.4] | 46.6 [6.0 to 81.9] | 50.1 [6.0 to 93.4]
  (90 days) Responders: number analyzed (Participants) | 5 | 4 | 9
  (90 days) Responders | 77.0 [53.4 to 99.8] | 62.1 [18.4 to 97.3] | 77.0 [18.4 to 99.8]
  (90 days) Nonresponders: number analyzed (Participants) | 4 | 2 | 6
  (90 days) Nonresponders | 39.1 [29.6 to 50.6] | 36.9 [6.0 to 67.8] | 39.1 [6.0 to 67.8]
  (180 days) Responders: number analyzed (Participants) | 5 | 2 | 7
  (180 days) Responders | 71.2 [29.6 to 99.8] | 57.8 [18.4 to 97.3] | 71.2 [18.4 to 99.8]
  (180 days) Nonresponders: number analyzed (Participants) | 4 | 2 | 6
  (180 days) Nonresponders | 47.6 [36.3 to 93.4] | 74.8 [67.8 to 81.9] | 60.6 [36.3 to 93.4]
Statistical Analysis 1: Comparison: Overall; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.020, Wilcoxon (Mann-Whitney) — Statistical significance defined as p <= 0.05. Data for 30 day timepoint
Statistical Analysis 2: Comparison: Overall; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.029, Wilcoxon (Mann-Whitney) — Statistical significance defined as p <= 0.05. Data for 90 day timepoint
Statistical Analysis 3: Comparison: Overall; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.94, Wilcoxon (Mann-Whitney) — Statistical significance defined as p <= 0.05. Data for 180 day timepoint

9. Secondary Outcome: Tumor Response by Quantitative European Association for the Study of the Liver (qEASL) Criteria
Description: Lipiodol deposition in the tumor will be measured using non contrast CT. The images from the non contrast CT will also be correlated with qEASL response separately using contrast CT, MRI and PET imaging. Response rates taken at 30 days, 90 days, 180 days. Per qEASL criteria:
  Complete Response (CR): Total disappearance of enhancing tumor volume in target lesions Partial Response (PR): At least 65% decrease in enhanced tumor volume after treatment.
  Overall Response: CR + PR
Time Frame: 6 months
Population: 16 HCC and 14 non-HCC subjects had complete data for qEASL analysis at 30day f/u, 9 HCC and 7 non-HCC at 90 day f/u, and 9 HCC and 5 non-HCC at 180 day f/u.
Measure: Count of Participants; unit: Participants
Arm/Group | Lipiodol (HCC) | Lipiodol (Non-HCC)
Number analyzed (Participants) | 16 | 14
Participants
  30 day f/u: Responders | 6 | 1
  30 day f/u: Non-responders | 10 | 13
  90 day f/u: number analyzed (Participants) | 9 | 7
  90 day f/u: Responders | 5 | 4
  90 day f/u: Non-responders | 4 | 3
  180 day f/u: number analyzed (Participants) | 9 | 5
  180 day f/u: Responders | 6 | 5
  180 day f/u: Non-responders | 3 | 0

10. Secondary Outcome: Baseline Enhancing Tumor and Response by qEASL Criteria
Description: Analysis of enhancing tumor (% of tumor that arterially enhances on MRI imaging) to correlate with responders/nonresponders by qEASL criteria. Responders are subjects that demonstrated Complete Response or Partial Response by qEASL criteria. Nonresponders are all other subjects.
Time Frame: 30 days, 90 days, 180 days
Population: as for outcome 2
Measure: Median (Full Range); unit: % tumor enhancement
Arm/Group | Lipiodol (HCC) | Lipiodol (Non-HCC) | Overall
Number analyzed (Participants) | 16 | 14 | 30
% tumor enhancement
  (30 day) Responders: number analyzed (Participants) | 6 | 1 | 7
  (30 day) Responders | 74.1 [50.6 to 97.6] | 81.9 [81.9 to 81.9] | 77.0 [50.6 to 97.6]
  (30 days) Nonresponders: number analyzed (Participants) | 10 | 13 | 23
  (30 days) Nonresponders | 46.0 [6.1 to 99.8] | 50.7 [6.0 to 97.3] | 50.1 [6.0 to 99.8]
  (90 days) Responders: number analyzed (Participants) | 5 | 3 | 8
  (90 days) Responders | 71.2 [50.6 to 99.8] | 81.9 [67.8 to 97.3] | 74.1 [50.6 to 99.8]
  (90 days) Nonresponders: number analyzed (Participants) | 4 | 3 | 7
  (90 days) Nonresponders | 39.1 [29.6 to 93.4] | 18.4 [6.0 to 42.4] | 36.3 [6.0 to 93.4]
  (180 days) Responders: number analyzed (Participants) | 6 | 4 | 10
  (180 days) Responders | 62.3 [29.6 to 99.8] | 74.8 [18.4 to 97.3] | 69.5 [18.4 to 99.8]
  (180 days) Nonresponders: number analyzed (Participants) | 3 | 0 | 3
  (180 days) Nonresponders | 41.8 [36.3 to 93.4] |  | 41.8 [36.3 to 93.4]
Statistical Analysis 1: Comparison: Overall; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.06, Wilcoxon (Mann-Whitney) — Statistical significance defined as p <= 0.05. Data for 30 day timepoint
Statistical Analysis 2: Comparison: Overall; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.013, Wilcoxon (Mann-Whitney) — Statistical significance defined as p <= 0.05. Data for 90 day timepoint
Statistical Analysis 3: Comparison: Overall; [analysis description as in outcome 2, analysis 1]; Test type: Other; p = 0.67, Wilcoxon (Mann-Whitney) — Statistical significance defined as p <= 0.05. Data for 180 day timepoint

11. Secondary Outcome: 6-month Survival Rate of Patients With HCC and Liver Metastases Treated With Conventional TACE
Description: Measure the association between baseline Lipiodol deposition and the 6-month survival rate by estimating median survival for each stratum, and by testing for homogeneity using a logrank test if hazards are proportional.
Time Frame: 6 months
Population: Kaplan-Meier survival analysis to estimate survival rate% at 6 months. Subjects are censored if survival is unknown at time point due to loss to followup.
Measure: Number; unit: percentage of partcipants
Arm/Group | Lipiodol
Number analyzed (Participants) | 39
percentage of partcipants | 67.6

ADVERSE EVENTS:
Time Frame: 6 months post treatment
Description: Adverse events determined by regular laboratory tests and clinical visits, reviewed by investigators.
Groups:
- Lipiodol/TACE: Lipiodol, 10cc per TACE.
  Lipiodol: Lipiodol is used as a carrier for chemotherapy agents and also as an occlusion agent. In TACE procedures, Lipiodol is mixed with the chemotherapy agent(s) and delivered to the tumor via the hepatic artery, causing necrosis of the targeted tumor(s).
  Adverse events assessed in relation to TACE procedure.
Arm/Group | Lipiodol/TACE
All-Cause Mortality (participants affected / at risk) | 2/39
Serious Adverse Events (participants affected / at risk) | 11/39
Other Adverse Events (participants affected / at risk) | 33/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lipiodol/TACE (N=39)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hepatic failure (Hepatobiliary disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Hepatic abscess (Gastrointestinal disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lipiodol/TACE (N=39)
Abdominal pain (Gastrointestinal disorders) | 4 (4)
Anemia (Blood and lymphatic system disorders) | 3 (4)
Ascites (Gastrointestinal disorders) | 2 (4)
Edema limbs (General disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 6 (7)
Alkaline phosphatase increased (Investigations) | 3 (3)
Aspartate aminotransferase (Investigations) | 9 (17)
Fatigue (General disorders) | 7 (9)
Fever (General disorders) | 2 (2)
Blood bilirubin increased (Investigations) | 3 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 3 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 (5)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Lymphocyte count decreased (Investigations) | 5 (6)
Nausea (Gastrointestinal disorders) | 6 (6)
Platelet count decreased (Investigations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2015-12-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT01877187/Prot_SAP_000.pdf
  • Informed Consent Form (2017-08-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT01877187/ICF_001.pdf